CLINICAL TRIAL: NCT01466881
Title: Phase II Trial of the Aurora Kinase A Inhibitor MLN8237, in Relapsed or Refractory Peripheral T-Cell Non-Hodgkin Lymphoma
Brief Title: Alisertib in Treating Patients With Relapsed or Refractory Peripheral T-Cell Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-03551; NCI-2011-03551 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SWOG-S1108; CDR0000714328; S1108 (Other: SWOG); S1108 (Other: CTEP); U10CA180888 (NIH); U10CA032102 (NIH)
Record Dates: First submitted 2011-11-03; First posted 2011-11-08 (Estimated); Results first posted 2016-03-10 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2015-01

CONDITIONS: Adult Nasal Type Extranodal NK/T-Cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-Cell Lymphoma; Hepatosplenic T-Cell Lymphoma; Mature T-Cell and NK-Cell Non-Hodgkin Lymphoma; Recurrent Adult Non-Hodgkin Lymphoma; Recurrent Adult T-Cell Leukemia/Lymphoma
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, T-Cell; Lymphoma, Non-Hodgkin; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — MLN 8237

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (alisertib) (Experimental): Patients receive alisertib PO BID on days 1-7. Treatment repeats every 21 days for 17 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Alisertib; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Alisertib — Given PO
  Other Names: Aurora A Kinase Inhibitor MLN8237; MLN-8237; MLN8237
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase II trial studies how well alisertib works in treating patients with peripheral T-cell non-Hodgkin lymphoma that has come back after a period of improvement or has not responded to treatment. Alisertib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the objective response rate (complete responses + partial responses) after treatment with alisertib (MLN8237) in patients with relapsed or refractory peripheral T-cell non-Hodgkin lymphoma.

II. To assess overall survival (OS) and progression-free survival (PFS) in this patient population.

III. To evaluate the safety and tolerability of MLN8237 treatment for this patient population.

IV. To explore the association between pre-treatment aurora kinase A expression in tumor biopsies as measured by fluorescence in situ hybridization (FISH) and objective response rate in patients with peripheral T-cell lymphomas (PTCL) treated with MLN8237.

IV. To investigate the copy number, mutational status, expression of aurora kinase (A, B, and C) and associated signaling pathways in PTCL utilizing tissue microarray analysis (TMA) before and after treatment with MLN8237.

V. To investigate changes in the serum cytokine profile pre- and post- aurora kinase Inhibitor treatment.

VI. To evaluate serum markers of apoptosis pre- and post- aurora kinase inhibitor treatment as pharmacodynamic markers of efficacy.

OUTLINE:

Patients receive alisertib orally (PO) twice daily (BID) on days 1-7. Treatment repeats every 21 days for 17 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 4 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed relapsed/refractory non-Hodgkin lymphoma (NHL) having progressed after a minimum of one systemic therapy with any of the following T-cell histologies:

  * Peripheral T-cell NHL (PTCL) not otherwise specified (NOS)
  * Anaplastic large cell T-cell lymphoma (ALCL) that is anaplastic lymphoma kinase either positive or negative
  * Angioimmunoblastic T-cell NHL
  * Subcutaneous panniculitis-like T-cell lymphoma
  * Enteropathy-associated T-cell NHL
  * Hepatosplenic T-cell lymphomas
  * Extranodal natural killer (NK)/T-cell lymphoma, nasal type
  * Adult T-cell leukemia/lymphoma
  * Unclassifiable PTCL
  * Transformed cutaneous T-cell lymphoma (CTCL) to PTCL with systemic involvement (not local skin transformation)
  * No other histologies are eligible; examples of ineligible histologies include: T-cell prolymphocytic leukemia, T-cell large granular lymphocytic leukemia, NK-cell leukemia, mycosis fungoides, Sezary syndrome, lymphomatoid papulosis, and primary CTCL
* Patients must have received at least one course of prior systemic therapy which may include chemotherapy, antibody therapy, or immunotherapy; for all forms of systemic therapy, patients must have completed therapy at least 21 days prior to registration; patients must not be within 84 days of radioimmunotherapy; steroids at a low dose for control of itching (up to the equivalent of 20 mg of prednisone daily) are allowed
* Patients may have received prior radiation in combination with systemic therapy; patients must not be within 21 days of external beam radiation therapy
* Patients must not have received a previous allogeneic stem cell transplant or be within 90 days of an autologous stem cell transplant
* Adequate sections and a paraffin block from the relapsed/refractory specimen must be submitted for review by the lymphoma pathology group; an adequate biopsy requires sufficient tissue to establish the architecture and a Revised European American Lymphoma (REAL) or World Health Organization (WHO) histologic subtype with certainty; thus, core biopsies, especially multiple core biopsies MAY be adequate; whereas, needle aspirations or cytologies are not adequate
* Patients must have bidimensionally measurable disease within 28 days prior to registration; a diagnostic quality computed tomography (CT) scan of the chest abdomen, pelvis, neck and positron emission tomography (PET)/CT must be performed within 28 days of registration (PET/CT scan can be done instead of separate PET and CT scans only if the CT component is a diagnostic CT with contrast); patients who also have non-measurable disease in addition to measurable disease must have all non-measurable disease assessed within 42 days prior to registration
* Patients must have a bilateral or unilateral bone marrow aspirate and biopsy performed within 42 days prior to registration
* Patients must not have clinical evidence of central nervous system involvement by lymphoma; any laboratory tests that are performed to assess clinical signs of central nervous system involvement must have been performed within 42 days prior to registration, and the results must be negative
* Patients must be able to swallow tablets
* Patients known to be human immunodeficiency virus (HIV)-positive must not have multi-drug resistant HIV infection, CD4 counts < 150/mcL, or other concurrent acquired immunodeficiency syndrome (AIDS)-defining conditions
* Patients must be offered the opportunity to consent to the banking of specimens for future use
* Absolute granulocyte count >= 1,500 cells/mcL; patients with documented marrow involvement may be transfused to this value
* Platelet count >= 75,000 cells/mcL; patients with documented marrow involvement may be transfused to this value
* Serum creatinine (mg/dL) =< institutional upper limit of normal (IULN) obtained within 14 days prior to registration
* Calculated creatinine clearance > 50 ml/min; the serum creatinine value used in the calculation must have been obtained within 14 days prior to registration
* Serum bilirubin =< 2 times institutional upper limit of normal
* Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) both =< 2.5 x IULN
* Serum lactate dehydrogenase (LDH) obtained within 14 days prior to registration
* Patients must have a Zubrod performance status of 0, 1, or 2
* Patients must NOT have New York Heart Association (NYHA) class II-IV heart failure
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for five years
* Pregnant or nursing women are not eligible; women/men of reproductive potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and for 4 months after completion of MLN8237 administration; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, the patient should inform the treating physician immediately
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-10; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Barr, Principal Investigator — SWOG Cancer Research Network
Locations (161):
- United States (160):
  - Providence Hospital, Mobile, Alabama
  - The University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - The University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - The University of Arizona Medical Center-University Campus, Tucson, Arizona
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills - Peninsula Hospitals, Burlingame, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Sutter Cancer Research Consortium, Novato, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Oncare Hawaii Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - OnCare Hawaii-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Oncare Hawaii Inc-Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Oncare Hawaii Inc-Pali Momi, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Hematology and Oncology Associates, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - North Shore Hematology Oncology, Libertyville, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Kansas City CCOP, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita CCOP, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Hematology/Oncology Clinic LLP, Baton Rouge, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center Shreveport, Shreveport, Louisiana
  - Union Hospital of Cecil County, Elkton MD, Maryland
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium CCOP, Ann Arbor, Michigan
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Metro-Minnesota NCI Community Oncology Research Program, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology and Hematology PA-Woodbury, Woodbury, Minnesota
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis University Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Montana Cancer Consortium CCOP, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Frontier Cancer Center and Blood Institute-Billings, Billings, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Laura and Issac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - University of Rochester, Rochester, New York
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - University of Cincinnati, Cincinnati, Ohio
  - Salem Hospital, Salem, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Roper Hospital, Charleston, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Audie L Murphy Veterans Affairs Hospital, San Antonio, Texas
  - Cancer Therapy and Research Center at The UT Health Science Center at San Antonio, San Antonio, Texas
  - University Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- BCCA-Vancouver Cancer Centre, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Barr PM, Li H, Spier C, Mahadevan D, LeBlanc M, Ul Haq M, Huber BD, Flowers CR, Wagner-Johnston ND, Horwitz SM, Fisher RI, Cheson BD, Smith SM, Kahl BS, Bartlett NL, Friedberg JW. Phase II Intergroup Trial of Alisertib in Relapsed and Refractory Peripheral T-Cell Lymphoma and Transformed Mycosis Fungoides: SWOG 1108. J Clin Oncol. 2015 Jul 20;33(21):2399-404. doi: 10.1200/JCO.2014.60.6327. Epub 2015 Jun 15. PMID 26077240

RESULTS

PARTICIPANT FLOW:
Groups:
- MLN8237: Patients receive MLN8237 (alisertib) PO BID on days 1-7. Treatment repeats every 21 days for 17 courses in the absence of disease progression or unacceptable toxicity
Period: Overall Study
Arm/Group | MLN8237
Started | 42
Eligible and Treated | 37
Completed | 2
Not Completed | 40
Not completed — Ineligible | 5
Not completed — Adverse Event | 6
Not completed — Progression/relapse | 20
Not completed — Death | 4
Not completed — Other reason not protocol specified | 5

BASELINE CHARACTERISTICS:
Population: Only eligible patients were included in the analysis.
Arm/Group | MLN8237
Number analyzed (Participants) | 37
Age, Continuous [Median (Full Range); unit: years] | 62.0 [21.6 to 86.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 24
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (Complete Responses (CR) + Partial Responses (PR))
Description: Objective disease status is evaluated according to the 2007 revised Cheson et al. criteria. Complete Response(CR) is a complete disappearance of all disease with the exception of nodes. No new lesions. previously enlarged organs must have regressed and not be palpable. Bone marrow (BM) must be negative if positive at baseline. Normalization of markers. Partial Response(PR) is a 50% decrease in the SPD for up to 6 identified dominant lesions, including spleenic and hepatic nodules from baseline. No new lesions and no increase in the size of liver, spleen or other nodes.
Time Frame: Up to 1 year after registration
Population: All eligible patients who started treatment were included in assessing response estimates.
Measure: Number; unit: participants
Arm/Group | MLN8237
Number analyzed (Participants) | 37
participants
  Complete Response | 2
  Partial Response | 7
  No response | 28

2. Secondary Outcome: Overall Survival (OS)
Description: Measure from date of registration to date of death due to any cause. Patients last known to be alive are censored at date of last contact.
Time Frame: Up to 2 years after registration
Population: Only eligible patients were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MLN8237
Number analyzed (Participants) | 37
Months | 8 [4.5 to 9.5]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Measured from date of registration to date of first observation of progressive disease or death due to any cause. Patients last known to be alive and without report of progressive disease are censored at date of last contact. Progressive disease is at least 50% increase in the sum of the product of the diameters (SPD) of target measurable nodal lesions over the smallest sum observed or ≥ 50% increase in the greatest transverse diameter (GTD) of any node > 1 cm in shortest axis, or ≥ 50% increase in the SPD of other target measurable lesions over the smallest sum observed. New bone marrow involvement. New lesion > 1.5 cm in longest axis, or ≥ 50% increase in GTD of any previously involved node with a diameter ≤ 1.0 cm in the short axis such that its longest axis is now > 1.5 cm. Lymph nodes with long axis is > 1.5 cm, or if the both the long and short axes are > 1 cm. PET should be positive if positive PET at baseline.
Time Frame: Up to 2 years after registration
Population: Only eligible patients were included in the analysis
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | MLN8237
Number analyzed (Participants) | 37
Months | 3 [2.2 to 4.3]

4. Secondary Outcome: To Evaluate the Safety and Tolerability of MLN8237 (Number of With Grade 3 Through Grade 5 Adverse Events That Are Related to MLN8237)
Description: Incidence of toxicity as assessed by the Common Terminology Criteria for Adverse Events version 4.0. For each patient, worst grade of each event type is reported. Grade 3 = Severe, Grade 4 = Life-threatening, Grade 5 = Fatal.
Time Frame: Up to 1 year after registration
Population: Eligible patients who had received any treatment were included in the adverse event summaries. Any CTCAE 4.0 event of Grade 3 (severe), Grade 4 (life threatening), or Grade 5 (fatal) which deemed to be related to protocol treatment are included.
Measure: Number; unit: Participants
Arm/Group | MLN8237
Number analyzed (Participants) | 37
Participants
  Abdominal pain | 1
  Alkaline phosphatase increased | 2
  Anemia | 12
  Anorexia | 1
  Back pain | 1
  Blood bilirubin increased | 1
  CD4 lymphocytes decreased | 2
  Diarrhea | 1
  Fatigue | 1
  Febrile neutropenia | 5
  Fever | 1
  Gastrointestinal disorders - Other, specify | 1
  Hypercalcemia | 1
  Hyperglycemia | 1
  Hypotension | 1
  Infections and infestations - Other, specify | 1
  Leukocytosis | 1
  Lung infection | 1
  Lymph gland infection | 1
  Lymphocyte count decreased | 8
  Mucositis oral | 4
  Neutrophil count decreased | 12
  Pain | 2
  Platelet count decreased | 9
  Rash maculo-papular | 2
  Sepsis | 1
  Skin and subcutaneous tissue disorders - Other | 1
  Skin infection | 1
  Toxic epidermal necrolysis | 1
  Treatment related secondary malignancy | 1
  White blood cell decreased | 7

5. Other Pre Specified Outcome: Aurora Kinase A Expression
Description: To explore the association between pre-treatment aurora kinase A expression in tumor biopsies as measured by fluorescence in situ hybridization (FISH) and objective response rate in patients with PTCL treated with MLN8237
Time Frame: Baseline
Population: Eligible patients who consented for correlative studies and had Aurora kinase A expression measured.
Measure: Mean (Standard Deviation); unit: proportion of positivity
Groups:
- Non-responders: Eligible patients who received protocol treatment and did not respond to the protocol treatment. Patients for whom response assessment was inadequate were considered non-responders.
- Responders: Eligible Patients who received protocol treatment and achieved complete or partial response.
Arm/Group | Non-responders | Responders
Number analyzed (Participants) | 19 | 3
proportion of positivity | 0.121 (0.096) | 0.063 (0.060)
Statistical Analysis 1: Comparison: Non-responders vs Responders; The null hypothesis is that there is no significant difference in Aurora kinase A expression between responders and non-responders; Test type: Superiority or Other; p = 0.2316, Wilcoxon (Mann-Whitney); Two-sided alpha level of 0.05

ADVERSE EVENTS:
Time Frame: Up to 1 year after registration
Description: Eligible patients who had received any treatment were included. Incidence of toxicity as assessed by the Common Terminology Criteria for Adverse Events version 4.0.
Arm/Group | MLN8237
Serious Adverse Events (participants affected / at risk) | 19/37
Other Adverse Events (participants affected / at risk) | 36/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MLN8237 (N=37)
Anemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Cardiac disorders-Other (Cardiac disorders) | 1
Heart failure (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Multi-organ failure (General disorders) | 1
Lung infection (Infections and infestations) | 1
Lymph gland infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Encephalopathy (Nervous system disorders) | 1
Facial nerve disorder (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Renal and urinary disorders-Other (Renal and urinary disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 2
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MLN8237 (N=37)
Anemia (Blood and lymphatic system disorders) | 23
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 4
Sinus tachycardia (Cardiac disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 8
Diarrhea (Gastrointestinal disorders) | 12
Dysphagia (Gastrointestinal disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 7
Oral pain (Gastrointestinal disorders) | 2
Rectal hemorrhage (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 6
Chills (General disorders) | 2
Edema limbs (General disorders) | 8
Fatigue (General disorders) | 23
Fever (General disorders) | 11
Pain (General disorders) | 9
Infections and infestations-Other (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
Skin infection (Infections and infestations) | 2
Upper respiratory infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 5
Alkaline phosphatase increased (Investigations) | 8
Aspartate aminotransferase increased (Investigations) | 7
Blood bilirubin increased (Investigations) | 4
CD4 lymphocytes decreased (Investigations) | 2
Creatinine increased (Investigations) | 7
Lymphocyte count decreased (Investigations) | 14
Neutrophil count decreased (Investigations) | 15
Platelet count decreased (Investigations) | 19
Weight loss (Investigations) | 4
White blood cell decreased (Investigations) | 15
Anorexia (Metabolism and nutrition disorders) | 8
Dehydration (Metabolism and nutrition disorders) | 4
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypernatremia (Metabolism and nutrition disorders) | 2
Hyperuricemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 9
Hypocalcemia (Metabolism and nutrition disorders) | 7
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 9
Back pain (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Headache (Nervous system disorders) | 4
Memory impairment (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 9
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 4
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2
Skin ulceration (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less